CLINICAL TRIAL: NCT01135901
Title: The VEND RISK-study. Preventing Diabetes Type 2 in Overweight Persons in the Værnes Region, Central-Norway.
Brief Title: Local Measures to Prevent Diabetes in the Værnes Region.
Acronym: VEND-RISK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2010/696-2
Record Dates: First submitted 2010-04-26; First posted 2010-06-03 (Estimated); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus Type 2; Obesity
Keywords: prevention; public health; community health services; Norway
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group programme (Experimental): Group based behaviour change programme
  Interventions: Behavioral: Behavioural change programme

INTERVENTIONS:
Behavioral: Behavioural change programme — The programme consists of a introductory course, organised physical activity 2-3 times a week, meetings every 3rd month with lectures and theme nights, and organising self-help groups.

SUMMARY:
This is a development project involving four different municipalities in Central Norway. The aim is to identify adults with overweight and with an increased risk of developing diabetes mellitus type 2, then to prevent the disease to develop by the means of a behaviour change programme. The programme is group based.

ELIGIBILITY:
Inclusion Criteria:

* Living in Central Norway
* Find Risc score > 15
* Written, informed consent

Exclusion Criteria:

* Severe mental disorder
* Not being able to function in the group programme

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Diabetes mellitus type 2 | Visit 1 (baseline) till Visit 9 (5 years)

CONTACTS AND LOCATIONS:
Overall Officials: Bård Kulseng, PhD, Principal Investigator — Norwegian University of Technology and Science
Locations (1):
- Vaernesregionen: Meraker, Stjørdal, Selbu, Tydal, Stjørdal, Norway

REFERENCES:
- [Result] Folling IS, Kulseng B, Midthjell K, Rangul V, Helvik AS. Individuals at high risk for type 2 diabetes invited to a lifestyle program: characteristics of participants versus non-participants (the HUNT Study) and 24-month follow-up of participants (the VEND-RISK Study). BMJ Open Diabetes Res Care. 2017 Jul 31;5(1):e000368. doi: 10.1136/bmjdrc-2016-000368. eCollection 2017. PMID 28878932
- [Derived] Folling IS, Klockner C, Devle MT, Kulseng B. Preventing type 2 diabetes, overweight and obesity in the Norwegian primary healthcare: a longitudinal design with 60 months follow-up results and a cross-sectional design with comparison of dropouts versus completers. BMJ Open. 2022 Mar 9;12(3):e054841. doi: 10.1136/bmjopen-2021-054841. PMID 35264353
- [Derived] Folling IS, Solbjor M, Midthjell K, Kulseng B, Helvik AS. Exploring lifestyle and risk in preventing type 2 diabetes-a nested qualitative study of older participants in a lifestyle intervention program (VEND-RISK). BMC Public Health. 2016 Aug 25;16(1):876. doi: 10.1186/s12889-016-3559-y. PMID 27557801